CLINICAL TRIAL: NCT01301326
Title: Pilot Randomized Clinical Trial Comparing Subthreshold Laser Treatment Versus Threshold Laser Treatment for Retinal Arterial Macroaneurysm
Brief Title: Subthreshold Laser Treatment Versus Threshold Laser Treatment for Symptomatic Retinal Arterial Macroaneurysm
Acronym: RAM-SUB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Francesco Bandello, Department of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAM-SUB
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-01

CONDITIONS: Aneurysm
Keywords: retinal arterial macroaneurysm; laser treatment
MeSH Terms: conditions — Aneurysm; Retinal Arterial Macroaneurysm | interventions — Speech Reception Threshold Test

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- subthreshold laser treatment (Experimental)
  Interventions: Device: subthreshold and threshold laser treatment
- threshold laser treatment (Active Comparator)
  Interventions: Device: Threshold laser treatment

INTERVENTIONS:
Device: subthreshold and threshold laser treatment — subthreshold laser treatment
  Other Names: subthreshold
  Arms: subthreshold laser treatment
Device: Threshold laser treatment — threshold laser treatment
  Other Names: threshold
  Arms: threshold laser treatment

SUMMARY:
Best treatment option of retinal arterial macroaneurysm is still controversial. A recent publication has shown that subthreshold laser treatment can be beneficial in improving visual acuity in eyes with symptomatic retinal arterial macroaneurysm. Aim of the study is to compare the effects of subthreshold laser treatment and threshold laser treatment in patients affected by symptomatic retinal arterial macroaneurysm.

DETAILED DESCRIPTION:
The treatment of RAM is controversial and at present there is no general consensus about the best approach. Spontaneous obliteration of RAM may occur over the follow-up, but the long persistence of blood or subretinal fluid may lead to progressive photoreceptor damage, with consequent irreversible visual impairment. More specifically, the presence of subretinal hemorrhage beneath the fovea leads to a diminished visual function.

Treatment is generally indicated for RAM associated with exudative manifestations involving the fovea which do not tend to resolve spontaneously. The most commonly employed approach is direct or indirect laser photocoagulation with visible end-point. Nevertheless, several complications may be associated with conventional threshold laser for macular lesions, including enlargement of laser scar, choroidal neovascularization, and subretinal fibrosis. In addition to these complications, arteriolar obliteration, increased retinal exudation and scarring, with possible retinal traction, have also been reported as possible sequelae of the laser photocoagulation of RAM.

Another approach for the treatment of RAM is based on the use of subthreshold laser treatment.

Subthreshold laser treatment has been proposed in an attempt to minimize the negative aspects of conventional grid laser photocoagulation and has achieved encouraging results, especially in macular oedema secondary to diabetic retinopathy, proliferative diabetic retinopathy, and branch retinal vein occlusion. The concept underlying the use of subthreshold laser treatment is to decrease the laser damage by reducing the duration of laser exposure and by using a subvisible clinical end point. A micropulse diode laser releases low energy micropulses in order to confine the energy to the RPE cells, with limited protein denaturation, avoiding lateral thermal spreading.

Aim of the study is to compare the effects of subthreshold laser treatment to those of threshold laser treatment in patients affected by symptomatic retinal arterial macroaneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Retinal arterial macroaneurysm, exudative manifestations involving the fovea (including: subretinal/intraretinal fluid, and/or hard exudates, and/or hemorrhages), best corrected visual acuity worse than 20/80 Snellen equivalent, corresponding to 0.6 LogMAR

Exclusion Criteria:

* previous treatments for retinal arterial macroaneurysm, any other ocular disease

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
change in central point thickness | 6 months

SECONDARY OUTCOMES:
change in visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandello, MD, Study Chair — Department of Ophthalmology
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

REFERENCES:
- [Background] Parodi MB, Iacono P, Ravalico G, Bandello F. Subthreshold laser treatment for retinal arterial macroaneurysm. Br J Ophthalmol. 2011 Apr;95(4):534-8. doi: 10.1136/bjo.2009.175547. Epub 2010 Oct 17. PMID 20956278
- [Derived] Battaglia Parodi M, Iacono P, Pierro L, Papayannis A, Kontadakis S, Bandello FM. Subthreshold laser treatment versus threshold laser treatment for symptomatic retinal arterial macroaneurysm. Invest Ophthalmol Vis Sci. 2012 Apr 2;53(4):1783-6. doi: 10.1167/iovs.11-8772. PMID 22395893